CLINICAL TRIAL: NCT00688987
Title: Cortisol, Central Obesity, and Insulin Resistance: Long Term Studies in Addison's Patients
Brief Title: The Hypothalamic-Pituitary-Adrenal (HPA) Axis as an Effector System in Weight Regulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Jonathan Q. Purnell, OHSU - The Center for the Study of Weight Regulation
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: eIRB 545; OCTRI #711
Record Dates: First submitted 2008-05-30; First posted 2008-06-03 (Estimated); Last update posted 2008-06-05 (Estimated); Status verified 2008-06

CONDITIONS: Obesity; Addison's Disease
MeSH Terms: conditions — Obesity; Addison Disease | interventions — Hydrocortisone

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Subjects with AI will be randomized to each of three doses of hydrocortisone for 4 months on each dose.
  Interventions: Drug: Hydrocortisone
- 2 (Active Comparator): isocaloric diet
  Interventions: Dietary Supplement: Isocaloric Diet

INTERVENTIONS:
Drug: Hydrocortisone — Subjects will receive in random order daily (split) dosing of hydrocortisone: a low dose of 15 mg (10 in AM, 5 in PM); a medium dose of 25 mg (15 in AM, 10 in PM) and high dose of 40 mg (30 in AM, 10 in PM) for 4 months.
  Arms: 1
Dietary Supplement: Isocaloric Diet — Subjects will eat an isocaloric diet for 4 weeks while taking hydrocortisone
  Other Names: Weight stable diet
  Arms: 2

SUMMARY:
Replacing glucocorticoid in a dose dependent manner (including doses within the physiological range) to subjects with adrenal insufficiency will increase visceral fat accumulation independently of total fat mass.

DETAILED DESCRIPTION:
To measure total fat mass by DEXA scan, central (visceral) fat accumulation, insulin sensitivity by FSIVGTT, lipid levels, and adipocyte gene expression in subjects with AI receiving increasing doses of hydrocortisone replacement (15 mg, 25 mg, and 40 mg per day in split doses) for 4-months at a time during ad-lib feeding.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with complete adrenal failure as defined as spontaneous serum cortisol of levels less than 5 g/dl after 12 hours without glucocorticoid replacement and peak serum cortisol of < 5 g/dl 60 minutes after a 250 g ACTH stimulation test.
* Subjects who are at their usual weight (weight stable for at least 1 year)
* Subjects on stable replacement doses of any required hormone such as thyroid, sex hormones, mineralocorticoid replacement, growth hormone, and hydrocortisone for at least 6 months, and 4) have a normal body weight (BMI 19-27 kg/m2).

Exclusion Criteria:

* Possible confounders on body weight and insulin resistance
* Age less than 18 to exclude those who might be experiencing alterations in cortisol production or weight as a result of adolescent growth.
* Subjects who exercise > 30 minutes/day, 3 times a week.
* Smokers.
* Heavy alcohol drinkers (> 2 drinks/ day).
* Subjects with medical diagnosis including diabetes, heart disease, and cancer.
* Subjects with psychiatric illness (i.e., depression, psychosis, bipolar, schizophrenia; or are taking medications for these disorders).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2000-08; Primary Completion 2004-07 (Actual); Study Completion 2004-08 (Actual)

PRIMARY OUTCOMES:
Amounts of intra-abdominal fat and total fat at the end of the treatment period for each cortisol dose. | After 4 months on each dose

SECONDARY OUTCOMES:
Fasting Lipid levels, fat mass by DEXA, post-heparin lipase activity, insulin sensitivity, and fat biopsy | After 4-months on each dose

CONTACTS AND LOCATIONS:
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States